CLINICAL TRIAL: NCT01584700
Title: Renal Artery Denervation in Chronic Heart Failure- Pilot
Brief Title: Renal Artery Denervation in Chronic Heart Failure
Acronym: REACH-Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JROSM0135
Record Dates: First submitted 2011-09-29; First posted 2012-04-25 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2012-07

CONDITIONS: Congestive Cardiac Failure
Keywords: NYHA class III or IV; Maximal medical therapy; Not eligible for CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Artery Denervation (Other): Ontervention
  Interventions: Procedure: Renal Artery Denervation

INTERVENTIONS:
Procedure: Renal Artery Denervation — Radiofrequency ablation of the renal artery sympathetic outflow tract.

SUMMARY:
Heart failure is a common condition with debilitating symptoms and a poor prognosis. Patients with heart failure have a massively overactive sympathetic nervous system which attempts to compensate for their poorly functioning heart. This ultimately has only detrimental effects.

One of the principle mediators for this sympathetic response is found in the nerve cells in the kidneys. Whilst a significant proportion of medications used to treat heart failure act on these harmful pathways, none target the kidney sympathetic-nerve cells specifically. Additionally, because of their multiple sites of action these drugs all have side effects.

A new procedure that has recently been developed for the treatment of high blood pressure is renal denervation. This involves inserting a small catheter through the femoral artery and passing it to the kidney artery under x-ray guidance. From there, using radiofrequency waves, the sympathetic nerves within the kidney can be destroyed.

The investigators anticipate that this procedure will have a significant positive effect on patients with heart failure and aim to perform a pilot safety study on 7 individuals with advanced heart failure to assess its safety and effectiveness. The investigators hypothesise that renal artery denervation will lead to significant clinical and biochemical improvements in patients with marked heart failure.

DETAILED DESCRIPTION:
One of the key physiological changes seen in heart failure patients is overactivity of the sympathetic nervous system. This is a homeostatic response produced by the body in an attempt to compensate for a poorly functioning heart and the resultant underperfused tissues. In acute heart failure this has a positive effect but in chronic heart failure, the long standing sympathetic overactivity causes multiple undesirable side effects including profound vasoconstriction, increased sodium reabsorption by the kidneys, renin release and decreased renal blood flow. Afferent and efferent sympathetic chains in the renal artery play an important role in the mediation of this response.

Current management of heart failure principally hinges on drugs that attempt to attenuate or interrupt this response via renin angiotensin system, adrenoreceptors or the renal tubules. These drugs have multiple side effects, partly because of their multiple sites of action. None directly target the sympathetic discharge at its source.

The development of renal artery denervation opens a unique opportunity for potentially longlasting relief of this intense renal sympathetic over-activity. The technique has a current role in the management of resistant hypertension where it has shown very favourable results with minimal side effects. The investigators envisage that this technique could also be highly beneficial to patients with heart failure by directly interrupting this sympathetic overactivity. This initial study involving 7 patients is a pilot safety study to assess this potential.

ELIGIBILITY:
Inclusion Criteria:

* congestive cardiac failure
* maximal medical therapy
* NYHA class III/IV

Exclusion Criteria:

* clinically unstable
* pre-existing renal disease
* unfavourable anatomy
* tortuous femoral anatomy
* unable to consent
* CRT present or eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 1 year
  To ensure that patients with heart failure are able to acceptably tolerate the procedure and its potential effect on haemodynamics.

SECONDARY OUTCOMES:
NYHA classification | 1 year
  To assess NYHA classification of dyspnoea
6 minute walk test | 1 year
  To assess impact on 6 minute walk test
Cardiopulmonary testing | 1 year
  To assess the impact on cardiopulmonary exercise testing
NT-proBNP | 1 year
  To assess the impact on NT-proBNP levels
Urinary excretion of renal hormones | 1 year
  To assess the impact on the urinary excretion of renal hormones

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Davies, PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Hammersmith Hospital, London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided
waiting

REFERENCES:
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Derived] Davies JE, Manisty CH, Petraco R, Barron AJ, Unsworth B, Mayet J, Hamady M, Hughes AD, Sever PS, Sobotka PA, Francis DP. First-in-man safety evaluation of renal denervation for chronic systolic heart failure: primary outcome from REACH-Pilot study. Int J Cardiol. 2013 Jan 20;162(3):189-92. doi: 10.1016/j.ijcard.2012.09.019. Epub 2012 Sep 29. PMID 23031283